CLINICAL TRIAL: NCT03414502
Title: Treatment of Rheumatoid Arthritis With Disease-modifying Antirheumatic Drugs (DMARDs): Predictors of Response
Brief Title: Treatment of Rheumatoid Arthritis With DMARDs: Predictors of Response
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0439-23-FB
Record Dates: First submitted 2014-01-02; First posted 2018-01-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate; DMARD
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Abatacept; Adalimumab; Azathioprine; baricitinib; Certolizumab Pegol; Etanercept; golimumab; Hydroxychloroquine; Infliximab; Leflunomide; Minocycline; Rituximab; sarilumab; Sulfasalazine; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (16):
- Methotrexate Therapy (Active Comparator): Participants will receive methotrexate therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Methotrexate
- Abatacept Therapy (Active Comparator): Participants will receive abatacept therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Abatacept
- Adalimumab Therapy (Active Comparator): Participants will receive adalimumab therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Adalimumab
- Azathioprine Therapy (Active Comparator): Participants will receive azathioprine therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Azathioprine
- Barcitinib Therapy (Active Comparator): Participants will receive barcitinib therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Baricitinib
- Certolizumab Therapy (Active Comparator): Participants will receive certolizumab therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Certolizumab
- Etanercept Therapy (Active Comparator): Participants will receive etanercept therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Etanercept
- Golimumab Therapy (Active Comparator): Participants will receive golimumab therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Golimumab
- Hydroxycholoroquine Therapy (Active Comparator): Participants will receive hydroxychloroquine therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Hydroxychloroquine
- Infliximab Therapy (Active Comparator): Participants will receive infliximab therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Infliximab
- Leflunomide Therapy (Active Comparator): Participants will receive leflunomide therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Leflunomide
- Minocycline Therapy (Active Comparator): Participants will receive minocycline therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Minocycline
- Rituximab Therapy (Active Comparator): Participants will receive rituximab therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Rituximab
- Sarilumab Therapy (Active Comparator): Participants will receive sarilumab therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Sarilumab
- Sulfasalazine Therapy (Active Comparator): Participants will receive sulfasalazine therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Sulfasalazine
- Tofacitinib Therapy (Active Comparator): Participants will receive tofacitinib therapy for rheumatoid arthritis (RA) treatment.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Methotrexate — Starting dose of Methotrexate of 15 mg once a week plus folic acid 1mg daily.
  Other Names: Methotrexate (MTX)
  Arms: Methotrexate Therapy
Drug: Abatacept — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Orencia
  Arms: Abatacept Therapy
Drug: Adalimumab — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Humira
  Arms: Adalimumab Therapy
Drug: Azathioprine — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Imuran
  Arms: Azathioprine Therapy
Drug: Baricitinib — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Olimuant
  Arms: Barcitinib Therapy
Drug: Certolizumab — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Cimzia
  Arms: Certolizumab Therapy
Drug: Etanercept — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Enbrel
  Arms: Etanercept Therapy
Drug: Golimumab — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Simponi
  Arms: Golimumab Therapy
Drug: Hydroxychloroquine — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Plaquenil
  Arms: Hydroxycholoroquine Therapy
Drug: Infliximab — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Remicade
  Arms: Infliximab Therapy
Drug: Leflunomide — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Arava
  Arms: Leflunomide Therapy
Drug: Minocycline — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Minocin
  Arms: Minocycline Therapy
Drug: Rituximab — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Rituxin
  Arms: Rituximab Therapy
Drug: Sarilumab — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Kevzara
  Arms: Sarilumab Therapy
Drug: Sulfasalazine — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Azulfidine
  Arms: Sulfasalazine Therapy
Drug: Tofacitinib — Starting dose may be adjusted as needed at investigator's discretion.
  Other Names: Xeljanz
  Arms: Tofacitinib Therapy

SUMMARY:
Rheumatoid arthritis (RA) is a common disease with approximately 1% prevalence. RA is also a chronic, progressive disease with no cure. Current treatment goals are to minimize pain, limit joint damage, and prevent loss of function. Drugs used to treat RA include non-steroidal anti-inflammatory drugs (NSAIDS), glucocorticoids, and disease-modifying anti-rheumatic drugs (DMARDs), including biologics. Methotrexate (MTX) is the DMARD of choice in the treatment of RA, because it has been shown to be both well-tolerated and effective in achieving clinical response and slowing radiographic progression of disease. However, this drug alone results in remissions in only a small subset of patients and reliable predictors of DMARD response have yet to be identified.

This study is open-label of 16-weeks duration to identify factors that help predict clinical responses to disease-modifying antirheumatic drugs (DMARD) therapies for rheumatoid arthritis (RA) participants. All participants will receive a starting dose of DMARD medication(s) which may be adjusted by the investigator as needed. If a participant becomes intolerant of a DMARD medication, the participant will be withdrawn at the discretion of the investigator. Necessary withdrawals prior to week 16 visits will be considered end of study. Otherwise, end of study data as well as study serum will be collected at week 16. A portion of the blood collected at baseline, week 8 and week 16 for the optional addendum portion of the study is for future research and will be utilized attempting to look to detect the generation of superoxide radicals. These radicals have been shown to be associated with inflammation and may correlate with the progression of RA, which if confirmed, should decrease the levels of these radicals signaling response to treatment.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a common disease with approximately 1% prevalence. RA is also a chronic, progressive disease with no cure. Current treatment goals are to minimize pain, limit joint damage, and prevent loss of function. Drugs used to treat RA include non-steroidal anti-inflammatory drugs (NSAIDS), glucocorticoids, and disease-modifying anti-rheumatic drugs (DMARDs), including biologics. Methotrexate (MTX) is the DMARD of choice in the treatment of RA, because it has been shown to be both well-tolerated and effective in achieving clinical response and slowing radiographic progression of disease. However, this drug alone results in remissions in only a small subset of patients and reliable predictors of DMARD response have yet to be identified.

Investigators have examined the discriminatory characteristics of several clinical and biologic parameters in predicting treatment response (at least 50% improvement based on American College of Rheumatology criteria), including rheumatoid factor (RF) isotypes (particularly Immunoglobulin A (IgA) and Immunoglobulin M (IgM), matrix metalloproteinase (MMP)-3, human leukocyte antigen-DR isotope (HLA-DRB1) shared epitope (SE)-containing alleles, C-reactive protein, and interleukin (IL)-1.

The purpose of the study is to prospectively gather information on participants with rheumatoid arthritis (RA) and their response to disease-modifying antirheumatic drugs (DMARD) therapy. Specifically, to evaluate the efficacy of DMARD therapy as defined by attaining American College of Rheumatology 50 (ACR50) response after 16 weeks of therapy and to identify predictors of DMARD response, such as genetic factors, serological factors or co-morbid conditions. A maximum of 400 rheumatoid arthritis (RA) participants will be enrolled in this 16-week, open-label study. Adult males and females will be enrolled, but RA is approximately three times more common in females.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosed rheumatoid arthritis (RA) with 4 of 7 American College of Rheumatology criteria

  * Morning stiffness for at least 1 hour for at least 6 weeks
  * Swelling of 3 or more joints for at least 6 weeks
  * Swelling of wrist, metacarpophalangeal (MCP), or proximal interphalangeal joints for 6 or more weeks
  * Symmetric joint swelling
  * Hand x-rays with erosions or bony decalcifications
  * RA nodules
  * Rheumatoid factor (RF) positive
* >19 yrs old at RA diagnosis
* Active disease with at least 1 swollen joint
* Starting new DMARD medication(s) (abatacept, adalimumab, azathioprine, barcitinib, certolizumab, etanercept, golimumab, hydroxychloroquine, infliximab, leflunomide, methotrexate, minocycline, rituximab, sarilumab, sulfasalazine, tofacitinib)
* If on other DMARDS, must be on stable dose for ≥ 6 wks
* If on glucocorticoids, must be on stable dose for 2 wks (< 10mg of Prednisone/day or equivalent)
* Able to adhere to study visit schedule: enrollment (8 wks & 16 wks +/- 2 wks)
* Hemoglobin (Hgb) > 9g/dl
* Platelets >100
* Creatinine <1.6
* Aspartate transferase (AST) or alanine aminotransferase (ALT) at or below 1.2 x upper limit
* Albumin up to 1.0 g/dL below lower limit of normal

EXCLUSION CRITERIA:

* Pregnant or breastfeeding women
* Men and women of child bearing potential unwilling to practice effective method of contraception

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-12-10 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Disease-modifying Antirheumatic Drugs Therapy for Rheumatoid Arthritis | 16 weeks
  The efficacy of the disease-modifying antirheumatic drugs (DMARD) in the study will be determined using the American College of Rheumatology 50 (ACR50). This is a composite measure defined as both improvement of 50% in the number of tender and number of swollen joints, and a 50% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).

SECONDARY OUTCOMES:
Genetic factors as Predictors of Disease-modifying Antirheumatic Drugs Response | 16 weeks
  Based on American College of Rheumatology 50 (ACR50) composite measure after 16 weeks of treatment, the number of participants will be determined that have genetic factors, such as the shared epitope, that demonstrate a 50% improvement in the number of tender and swollen joints, and a 50% improvement in three of five criteria: patient global assessment, physician global assessment, functional ability measure (most often Health Assessment Questionnaire/HAQ), visual analog pain scale and erythrocyte sedimentation rate or C-reactive protein (CRP).
Serological Factors as Predictors of Disease-modifying Antirheumatic Drugs Response | 16 weeks
  Based on American College of Rheumatology 50 (ACR50) composite measure after 16 weeks of treatment, the number of participants will be determined that have serological factors, such as cyclic citrullinated peptide (CCP) isotypes, that demonstrate a 50% improvement in the number of tender and swollen joints, and a 50% improvement in three of five criteria: patient global assessment, physician global assessment, functional ability measure (most often Health Assessment Questionnaire/HAQ), visual analog pain scale and erythrocyte sedimentation rate or C-reactive protein (CRP).
Co-morbid Conditions as Predictors of Disease-modifying Antirheumatic Drugs Response | 16 weeks
  Based on American College of Rheumatology 50 (ACR50) composite measure after 16 weeks of treatment, the number of participants will be determined that have co-morbid conditions, such as periodontal disease, that demonstrate a 50% improvement in the number of tender and swollen joints, and a 50% improvement in three of five criteria: patient global assessment, physician global assessment, functional ability measure (most often Health Assessment Questionnaire/HAQ), visual analog pain scale and erythrocyte sedimentation rate or C-reactive protein (CRP).

CONTACTS AND LOCATIONS:
Overall Officials: James R O'Dell, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No